CLINICAL TRIAL: NCT07283588
Title: Intensive Care Burden of Sepsis in Türkiye: Analysis of Multicenter Two-time Point Prevalence Approach and Clinical Outcomes (İntensive Care Sepsis Prevelance in Turkey (INSEP-TURK))
Brief Title: İntensive Care Sepsis Prevelance in Turkey (INSEP-TURK)
Acronym: INSEP-TURK
Status: Active, not recruiting | Type: Observational
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mete Erdemir, study director, Gulhane Training and Research Hospital
Other Study IDs: 2025-354
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Septic Shock Point Prevalence; Sepsis
Keywords: Prevalence of Septic Shock; TÜRKİYE; POINT PREVALENCE; sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days

SUMMARY:
Sepsis is a life-threatening condition characterized by a dysregulated host response to infection, leading to tissue damage, multiple organ dysfunction (MODS), disseminated intravascular coagulation (DIC), and high mortality. Despite its global significance, robust epidemiological data from low- and middle-income countries, including Turkey, remain limited. This multicenter, two-timepoint point-prevalence study aims to determine the prevalence of sepsis and septic shock in adult intensive care units (ICUs) across Turkey and to evaluate associated clinical outcomes.The study will be conducted between September 2025 and January 2026 in adult ICUs nationwide. Sepsis and septic shock will be defined according to the 2021 Surviving Sepsis Campaign Guidelines. Detailed data will be collected on participating ICUs, clinicians, patient demographics, comorbidities, infection characteristics, organ dysfunction, laboratory findings, and treatments. Patients will be followed for 30 days to assess ICU length of stay, discharge status, mortality, and ventilator- and vasopressor-free days.The primary objective is to determine the point prevalence of sepsis and septic shock in Turkish ICUs. The secondary objective is to evaluate 30-day mortality among patients with sepsis and septic shock. The findings are expected to provide crucial epidemiological insights and help improve sepsis management strategies in Turkey.

DETAILED DESCRIPTION:
Sepsis is a systemic inflammatory response to infection that results in tissue injury, multiple organ dysfunction (MODS), disseminated intravascular coagulation (DIC), and dysregulation of the immune system through the activation of various toxic mediators. The exaggerated and dysregulated host response to infection constitutes the fundamental pathophysiological mechanism of sepsis and septic shock. According to data from the United States (USA) between 2004 and 2009, the incidence of sepsis was reported to be 300-1,031 per 100,000 population per year. During the same period, the mortality rate among patients diagnosed with sepsis was documented to be 15-30%. Studies conducted between 1979 and 2015 across seven high-income countries reported an incidence of severe sepsis of 270 per 100,000 population per year with a mortality rate of 26%. Sepsis and septic shock account for a substantial portion of healthcare expenditures worldwide. According to U.S. data from 2011, patients diagnosed with sepsis accounted for 6.2% of all hospital expenditures (23.7 million USD). The World Health Organization (WHO) declared improved prevention, recognition, and treatment of sepsis a global health priority in 2017.Septic shock is a condition associated with high mortality and morbidity. Survivors of sepsis are at increased risk for recurrent infections, repeated hospitalizations, reduced quality of life, and long-term mortality. Given the high morbidity and mortality associated with sepsis, early treatment before irreversible organ dysfunction develops is critically important. Large-scale epidemiological studies on sepsis remain limited in low- and middle-income countries, where approximately two-thirds of the world's population resides. The prevalence and mortality rates of sepsis in Turkey are largely unknown. Turkey is a middle-income country and is among the nations with high levels of antimicrobial resistance.Whether antimicrobial resistance alone increases mortality remains unclear. Previous studies have reported that infections caused by antibiotic-resistant bacteria are associated with higher mortality, longer ICU stays, and increased hospitalization costs. This study was designed as a multicenter, two-timepoint investigation to assess the prevalence of sepsis in intensive care units across Turkey and evaluate associated clinical outcomes.Materials and MethodsA multicenter, two-timepoint (September 2025-January 2026), point-prevalence and clinical outcome analysis will be conducted across Turkey on dates determined by the study coordinator. Informed consent will be obtained from all participating patients. Data from participating centers will be collected electronically or in written form.Definitions of sepsis and septic shock will follow the 2021 Surviving Sepsis Campaign Guidelines (SSCG). Sepsis will be defined as clinically suspected infection together with at least one organ dysfunction, indicated by an increase of ≥2 points in the SOFA score. Septic shock will be defined as persistent hypotension requiring vasopressor therapy despite adequate fluid resuscitation and a serum lactate level >2 mmol/L.Information regarding the participating ICUs will include the hospital name, institutional affiliation, clinical experience of ICU physicians, physician specialty, ICU service type, ICU level, number of ICU beds, total number of patients with sepsis and septic shock on the study day, and patient-to-physician ratio.Patient-level data will include demographics and comorbidities: age, sex, ICU day on the study date, admission source, primary diagnosis, APACHE II score on admission, SOFA score on the study day, and treatments received within the 24 hours preceding the study day (vasoactive therapies, corticosteroids, albumin, blood transfusions, IVIG, renal replacement therapy, plasma exchange/plasmapheresis, cytokine adsorption, ECMO, mechanical ventilation). Additional information will include the use and duration of corticosteroid therapy, infection focus (urinary tract, lower respiratory tract, bloodstream, intra-abdominal, genitourinary, central nervous system, soft tissue, surgical site), infection type (hospital-acquired or community-acquired), presence of multiple infection sites, polymicrobial infection status, pathogen class (Gram-positive bacteria, Gram-negative bacteria, fungi, viruses, unidentified), pathogen species, antibiotic regimen used for sepsis, and presence of septic shock on the study day.Comorbidities will include: solid organ malignancies, insulin-dependent diabetes mellitus, cerebrovascular disease, New York Heart Association (NYHA) class III-IV heart failure, COPD, restrictive or vascular pulmonary disease, chronic liver failure, chronic renal failure (creatinine ≥2 mg/dL or dialysis), and immunosuppression. Immunosuppression will be defined as neutropenia (<500 mm-3), hematologic malignancy, splenectomy, HIV infection, chemotherapy or radiotherapy within 6 months prior to ICU admission, corticosteroid therapy prior to ICU admission (prednisolone >40 mg/day, hydrocortisone >160 mg/day, methylprednisolone >32 mg/day, dexamethasone >6 mg/day for >2 weeks), post-transplantation status, or chronic alcoholism.Laboratory data will include: highest WBC count (mm³), lowest platelet count (mm³), highest ALT (U/L), highest lactate (mmol/L), highest CRP (mg/dL), highest creatinine (mg/dL), highest BUN (mg/dL), highest total bilirubin (mg/dL), highest INR, highest procalcitonin (ng/mL), lowest albumin (g/dL), lowest PaO₂/FiO₂ ratio, and lowest ScvO₂ on the study day. Sepsis-related organ dysfunctions (cardiovascular, respiratory, renal, hepatic, hematologic, neurological) will also be recorded.On day 30 following the study date, the following outcomes will be assessed: ICU length of stay, ICU discharge status (discharged, transferred to ward, deceased), 30-day mortality, ventilator-free days, and vasopressor/inotrope-free days.Community-acquired infection will be defined as infection detected within the first 48 hours of ICU admission. Hospital-acquired infection will be defined as infection detected >48 hours after ICU admission.Primary OutcomeTo determine the point prevalence of sepsis and septic shock in intensive care units across Turkey on the study day.Secondary OutcomeTo evaluate 30-day mortality among patients diagnosed with sepsis and septic shock.Study Population / SampleThe study will be conducted in adult ICUs across Turkey that provide care to patients aged >18 years.LimitationsAs an observational study, randomization cannot be performed. Additionally, variations in clinical practice, resource availability, and patient characteristics across participating ICUs may limit generalizability.HypothesesH0:The prevalence of sepsis and septic shock in adult ICUs across Turkey is low and does not significantly influence clinical outcomes.H1:The prevalence of sepsis and septic shock in adult ICUs across Turkey is high and exerts a significant impact on clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* The study will be conducted in adult intensive care units across Turkey, including patients aged 18 years and older.

Exclusion Criteria:

* Individuals under 18 years of age
* Individuals who do not consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in adult intensive care units across Turkey, including patients aged 18 years and older.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Point-prevalence of sepsis and septic shock in adult ICU patients in Turkey | On the study day (two time points: September 2025 and January 2026)
  The proportion of adult patients in participating ICUs who meet the 2021 Surviving Sepsis Campaign criteria for sepsis or septic shock on the study day.

SECONDARY OUTCOMES:
30-day mortality among ICU patients with sepsis or septic shock | 30 days post-study day
  Mortality status at 30 days after the study day, including ICU discharge, transfer, or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Hylander Moller M, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock 2021. Crit Care Med. 2021 Nov 1;49(11):e1063-e1143. doi: 10.1097/CCM.0000000000005337. No abstract available. PMID 34605781
- [Result] Fleischmann-Struzek C, Mellhammar L, Rose N, Cassini A, Rudd KE, Schlattmann P, Allegranzi B, Reinhart K. Incidence and mortality of hospital- and ICU-treated sepsis: results from an updated and expanded systematic review and meta-analysis. Intensive Care Med. 2020 Aug;46(8):1552-1562. doi: 10.1007/s00134-020-06151-x. Epub 2020 Jun 22. PMID 32572531
- [Result] Connelly-Smith L, Alquist CR, Aqui NA, Hofmann JC, Klingel R, Onwuemene OA, Patriquin CJ, Pham HP, Sanchez AP, Schneiderman J, Witt V, Zantek ND, Dunbar NM. Guidelines on the Use of Therapeutic Apheresis in Clinical Practice - Evidence-Based Approach from the Writing Committee of the American Society for Apheresis: The Ninth Special Issue. J Clin Apher. 2023 Apr;38(2):77-278. doi: 10.1002/jca.22043. PMID 37017433
- [Result] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338